CLINICAL TRIAL: NCT04542317
Title: Cluster Randomized Controlled Trial to Test the Efficacy of a Psychosocial Intervention (REACH VN) to Support Alzheimer's Family Caregivers in Vietnam
Brief Title: Efficacy of a Dementia Family Caregiver Support Intervention in Vietnam
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Geriatric Hospital (Other Government); University of Minnesota (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1574137; R01AG064688 (NIH); TR001860 (Other Grant/Funding Number: National Center for Advancing Translational Sciences)
Record Dates: First submitted 2020-08-31; First posted 2020-09-09 (Actual); Results first posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Dementia
Keywords: Family caregiving
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: The active treatment is REACH VN, a culturally adapted version of REACH VA, a multi-component dementia family caregiver support intervention that includes psychoeducation, stress reduction, problem-solving, and skill-building.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REACH VN (Experimental): A multi-component behavioral intervention to support family caregivers of persons with dementia. Participants will receive 4-6 sessions in-person or by phone over the course of 2-3 months.
  Interventions: Behavioral: REACH VN
- Enhanced control (Placebo Comparator): A single session focused on education about the nature of dementia.
  Interventions: Behavioral: Enhanced control

INTERVENTIONS:
Behavioral: REACH VN — 4-6 sessions delivered over the course of 2-3 months.
  Arms: REACH VN
Behavioral: Enhanced control — A single session providing education about dementia
  Arms: Enhanced control

SUMMARY:
This is a cluster randomized controlled trial to test the efficacy of a psychosocial intervention to support family caregivers of persons living with dementia in Vietnam.

DETAILED DESCRIPTION:
The objective of this study is to conduct a cluster randomized controlled trial (RCT) to test the efficacy of a psychosocial intervention to support Alzheimer's family caregivers in Vietnam. The cluster RCT will test the hypothesis that family caregivers who receive the intervention will show lower psychological distress and lower caregiver burden compared with those in the control group (primary outcomes). In addition, we will conduct secondary analyses to examine whether the intervention group has lower perceived stress and somatic symptoms. Exploratory analyses will be conducted to determine if intervention effects are mediated by caregiver self-efficacy or knowledge gain.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for the cluster RCT, the family member will need to be the identified adult (age 18 and above) primary caregiver (i.e. the person spending who provides the most time day-to-day providing care) to an older adult with dementia who is living in the community. In the event that the primary caregiver is not available to participate, an alternate family member who provides substantial care (i.e., at least 4 hours/day) to the older adult with dementia will be eligible.
* Caregivers will need to score ≥ 6 on the Zarit Burden Inventory 4-item version.
* All participants will be living in designated clusters in Hai Duong, Vietnam.
* To be eligible, clusters will have a minimum of 5 participants and a maximum of 15 participants. Clusters will be defined as geographic areas serving local health stations.

Exclusion Criteria:

- Significant cognitive impairment or sensory deficit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Based on self-representation of gender identity.
Enrollment: 350 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-02-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vietnam National Geriatric Hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tran D, Nguyen H, Pham T, Nguyen AT, Nguyen HT, Nguyen NB, Nguyen BH, Harvey D, Gitlin L, Hinton L. Resources for Enhancing Alzheimer's Caregiver Health in Vietnam (REACH VN): study protocol for a cluster randomized controlled trial to test the efficacy of a family dementia caregiver intervention in Vietnam. Trials. 2022 May 9;23(1):377. doi: 10.1186/s13063-022-06228-6. PMID 35534904

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 41 clusters were randomized. 20 clusters were allocated to enhanced control, and 21 clusters were allocated to REACH VN intervention. 306 caregivers in enhanced control arm and 354 caregivers in REACH VN arm were assess for eligibility. During the subsequent screening process, we excluded one control cluster because the number of enrolled caregivers was below the threshold of five, leaving 40 enrolled clusters at the start of the study (21 intervention and 19 enhanced control).
Units Other Than Participants: cluster
Period: Overall Study
Arm/Group | REACH VN | Enhanced Control
Started | 175; 21 cluster | 175; 19 cluster
Completed | 148; 21 cluster | 157; 19 cluster
Not Completed | 27; 0 cluster | 18; 0 cluster
Not completed — Care recipients passed away | 18 | 13
Not completed — No longer a primary caregiver | 5 | 1
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Caregivers passed away | 0 | 2

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are reported only for participants who completed the 3-month follow-up. Participants who dropped out before the 3-month follow-up are not included in the baseline analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | REACH VN | Enhanced Control | Total
Number analyzed (Participants) | 160 | 170 | 330
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (10.9) | 61.4 (11.3) | 61.7 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116 | 117 | 233
  Male | 44 | 53 | 97
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 160 | 170 | 330
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 160 | 170 | 330
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Zarit Burden Interview-12 (ZBI-12) [Mean (Standard Deviation); unit: score on a scale] — The Zarit Burden Interview-12 (ZBI-12) asked caregivers to rate on a scale of 0 (never) to 4 (nearly always) how often they have experienced feelings of burden or stress related to caregiving (total score range: 0-48). A higher score indicates a higher feel of burden.
  score on a scale | 21.4 (8.4) | 22.0 (8.6) | 21.7 (8.5)
Patient Health Questionnaire-4 (PHQ-4) [Mean (Standard Deviation); unit: score on a scale] — Patient Health Questionnaire-4 (PHQ-4) asked caregivers to rate on a scale of 0 (not at all) to 3 (nearly every day) how often they have been bothered by symptoms (e.g., feeling nervous, anxious, or on edge) over the past two weeks (total score range: 0-12). A higher score indicates a higher severity.
  score on a scale | 3.7 (3.4) | 3.8 (3.6) | 3.7 (3.5)
Perceived Stress Scale (PSS-10) [Mean (Standard Deviation); unit: score on a scale] — In the Perceived Stress Scale-10 (PSS-10), caregivers were asked to rate on a scale of 0 (never) to 4 (very often) how often they have felt a certain way (e.g., been upset because of something that happened unexpectedly) within the past month (total score range: 0-40). A higher sore indicates a higher perceived stress.
  score on a scale | 13.7 (6.8) | 14.1 (6.7) | 13.9 (6.75)
Patient Health Questionnaire-15 (PHQ-15) [Mean (Standard Deviation); unit: score on a scale] — In the Patient Health Questionnaire-15 (PHQ-15), caregivers were asked to rate on a 3-point scale (0 = not bothered at all, 1 = bothered a little, 2 = bothered a lot) how much they have been bothered by somatic symptoms (e.g., stomach pain, headaches) during the past seven days (total score range: 0-30). A higher scores indicate a greater severity.
  score on a scale | 9.0 (5.4) | 9.0 (5.2) | 9.0 (5.3)

OUTCOME MEASURES:

1. Primary Outcome: Zarit Burden Interview-12 (ZBI-12)
Description: The Zarit Burden Interview-12 (ZBI-12) asked caregivers to rate on a scale of 0 (never) to 4 (nearly always) how often they have experienced feelings of burden or stress related to caregiving (total score range: 0-48). A higher score indicates a higher feel of burden.
Time Frame: Baseline period at month 0, follow up period at 3 months, and follow up period at 6 months
Population: The analytic sample included participants who completed at least 3-month assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | REACH VN | Enhanced Control
Number analyzed (Participants) | 160 | 170
score on a scale
  Baseline | 21.4 (8.4) | 22.0 (6.8)
  3 months | 20.1 (8.8) | 22.3 (8.8)
  6 months: number analyzed (Participants) | 148 | 157
  6 months | 19.2 (9.1) | 22.4 (8.6)

2. Primary Outcome: Patient Health Questionnaire-4 (PHQ-4)
Description: Patient Health Questionnaire-4 (PHQ-4) asked caregivers to rate on a scale of 0 (not at all) to 3 (nearly every day) how often they have been bothered by symptoms (e.g., feeling nervous, anxious, or on edge) over the past two weeks (total score range: 0-12). A higher score indicates a higher severity.
Time Frame: Baseline period at month 0, follow up period at 3 months, and follow up period at 6 months
Population: The analytic sample included participants who completed at least 3-month assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | REACH VN | Enhanced Control
Number analyzed (Participants) | 160 | 170
score on a scale
  Baseline | 3.7 (3.4) | 3.8 (3.6)
  3 months | 2.9 (3.0) | 4.4 (3.7)
  6 months: number analyzed (Participants) | 148 | 157
  6 months | 3.4 (3.3) | 3.8 (3.2)

3. Secondary Outcome: Perceived Stress Scale (PSS-10)
Description: In the Perceived Stress Scale-10 (PSS-10), caregivers were asked to rate on a scale of 0 (never) to 4 (very often) how often they have felt a certain way (e.g., been upset because of something that happened unexpectedly) within the past month (total score range: 0-40). A higher sore indicates a higher perceived stress.
Time Frame: Baseline period at month 0, follow up period at 3 months, and follow up period at 6 months
Population: The analytic sample included participants who completed at least 3-month assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | REACH VN | Enhanced Control
Number analyzed (Participants) | 160 | 170
score on a scale
  Baseline | 13.7 (6.8) | 14.1 (6.7)
  3 months | 11.9 (6.9) | 14.1 (6.7)
  6 months: number analyzed (Participants) | 148 | 157
  6 months | 12.7 (7.2) | 13.7 (6.8)

4. Secondary Outcome: Patient Health Questionnaire-15 (PHQ-15)
Description: In the Patient Health Questionnaire-15 (PHQ-15), caregivers were asked to rate on a 3-point scale (0 = not bothered at all, 1 = bothered a little, 2 = bothered a lot) how much they have been bothered by somatic symptoms (e.g., stomach pain, headaches) during the past seven days (total score range: 0-30). A higher score indicates a greater severity.
Time Frame: Baseline period at month 0, follow up period at 3 months, and follow up period at 6 months
Population: The analytic sample included participants who completed at least 3-month assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | REACH VN | Enhanced Control
Number analyzed (Participants) | 160 | 170
score on a scale
  Baseline | 9.0 (5.4) | 9.0 (5.2)
  3 months | 7.6 (4.5) | 9.5 (5.7)
  6 months: number analyzed (Participants) | 148 | 157
  6 months | 8.2 (5.1) | 8.8 (5.1)

ADVERSE EVENTS:
Time Frame: For each participant, adverse events were collected for the duration of participation in the study (up to 6 months)
Arm/Group | REACH VN | Enhanced Control
All-Cause Mortality (participants affected / at risk) | 0/175 | 2/175
Serious Adverse Events (participants affected / at risk) | 0/175 | 0/175
Other Adverse Events (participants affected / at risk) | 0/175 | 0/175

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-05-23): https://cdn.clinicaltrials.gov/large-docs/17/NCT04542317/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-15): https://cdn.clinicaltrials.gov/large-docs/17/NCT04542317/SAP_001.pdf
  • Informed Consent Form (2020-07-26): https://cdn.clinicaltrials.gov/large-docs/17/NCT04542317/ICF_002.pdf